CLINICAL TRIAL: NCT01561157
Title: Longitudinal Study of the Porphyrias
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Manisha C Balwani, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 10-1102; U54DK083909 (NIH)
Record Dates: First submitted 2012-02-13; First posted 2012-03-22 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Porphyrias; Cutaneous Porphyrias
Keywords: porphyria; acute intermittent; coproporphyria; variegate; erythropoietic; protoporphyria; hepatoerythropoietic; cutanea tarda; AIP; HCP; VP; ADP; ALAD; PCT; HEP; CEP; EPP; XLP; homozygous dominant; acute hepatic; AHP
MeSH Terms: conditions — Porphyria, Acute Intermittent; Porphyrias; Coproporphyria; Protoporphyria, Erythropoietic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood, plasma/serum, red blood cells, urine, tissue, DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (10):
- Acute Intermittent Porphyria (AIP): Patients with a documented diagnosis of AIP
- Hereditary Coproporphyria (HCP): Patients with a documented diagnosis of HCP
- Variegate Porphyria (VP): Patients with a documented diagnosis of VP
- Congenital Erythropoietic Porphyria (CEP): Patients with a documented diagnosis of CEP
- Hepatoerythropoietic Porphyria (HEP): Patients with a documented diagnosis of HEP
- Porphyria Cutanea Tarda (PCT): Patients with a documented diagnosis of PCT
- Erythropoietic Protoporphyria (EPP): Patients with a documented diagnosis of EPP
- X-Linked Protoporphyria (XLP): Patients with a documented diagnosis of XLP
- Aminolevulinate-Dehydratase Deficiency Porphyria (ALAD, ADP): Patients with a documented diagnosis of ALAD, ADP
- Homozygous Dominant Acute Hepatic Porphyria: Patients with a documented diagnosis of Homozygous Dominant AHP

SUMMARY:
The objective of this protocol is to conduct a longitudinal multidisciplinary investigation of the human porphyrias including the natural history, morbidity, pregnancy outcomes, and mortality in people with these disorders.

DETAILED DESCRIPTION:
The porphyrias are a group of rare metabolic diseases that may present in childhood or adult life and are due to deficiencies of enzymes in the heme biosynthetic pathway. The most common manifestations are related to accumulation of intermediates in the pathway and usually occur as acute neurological attacks, or cutaneous photosensitivity. Multiple mutations have been identified in each of the porphyrias. The risk of disability or death from these disorders is significant, in part because diagnosis is often delayed due to lack of adoption of diagnostic testing in clinical practice. Moreover, the natural history of these disorders is not well described and it is not known what determines differences in outcomes. New therapies are needed. For existing therapies, high-quality evidence on short and long term efficacy and safety is generally lacking. Therefore, the purpose of this long-term follow-up study of a large group of patients with the various porphyrias is to provide a better understanding of the natural history of these disorders, as affected by available therapies, and to aid in developing new forms of treatment.

The Office of Rare Diseases (ORD) of the National Institutes of Health (NIH) established a Rare Diseases Clinical Research Network (RDCRN) in collaboration with other NIH Institutes and currently has funded several rare diseases clinical research consortia and one Data Management and Coordinating Center. The Porphyrias Consortium was created as part of the RDCRN, to study the human porphyrias. The Porphyrias Consortium is a consortium of the academic institutions listed in the participating institutions table. All Centers in the Porphyrias Consortium are participating in the Longitudinal Study of the Porphyrias. Additional centers may be added if funding is available.

The initial objective of this protocol is to assemble a well-documented group of patients with confirmed diagnoses of specific porphyrias for clinical, biochemical, and genetic studies. The long-term objective is to conduct a longitudinal investigation of the natural history, complications, and therapeutic outcomes in people with acute and cutaneous porphyria.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a documented diagnosis of a porphyria.
* For each type of porphyria, the inclusion criteria are based on

  * Biochemical findings, as documented by laboratory reports (or copies) of porphyria-specific testing performed after 1980 (Absolute values are preferred for diagnostic biochemical thresholds. Fold increases in comparison to an upper (or lower) limit of normal (ULN or LLN) are also acceptable, but are complicated by considerable variation between laboratories in normal limits. Equivocal biochemical measurements may require confirmation by a consortium reference laboratory;)
  * molecular findings documenting the identification of a mutation in a porphyria-related gene.
* In addition, an individual or a parent or guardian must be willing to give written informed consent or assent, as appropriate.
* Provision is made for enrolling relatives who may not have symptoms but have biochemical or molecular documentation of a porphyria, or in the case of recessive disorders carry a disease-related mutation.

Exclusion Criteria:

* Cases with elevations of porphyrins in urine, plasma or erythrocytes due to other diseases (i.e. secondary porphyrinuria or porphyrinemia), such as liver and bone marrow diseases;
* Patients with a prior diagnosis of porphyria that cannot be documented by review of existing medical records or repeat biochemical or DNA testing.

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the following resources:
  1. Patients followed by one of the Investigators
  2. United Porphyrias Association (UPA)
  3. Non-study Physician referrals
  4. Self-referrals, including family members of individuals diagnosed with Porphyria (proband) and other individuals who may have heard about the study from other subjects or prospective subjects.
  5. Medical Records Review
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-11-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
clinical analysis | baseline
  To develop disease severity scores to describe the combined frequency and severity of disease manifestations, utilizing linear mixed effects models & stratification by age of onset.
Laboratory analysis | baseline
  To evaluate porphyrin and porphyrin precursor levels alone or by genotype and porphyria subtype

SECONDARY OUTCOMES:
Relationship between disease severity and biomarkers | baseline
  To develop longitudinal models that relate, for example, porphyrin and porphyrin precursor levels alone or in concert with age, genotype and other features to the disease manifestation frequency.
Effectiveness and tolerability of currently used and new therapies for the human porphyrias | baseline
  Qualitative evaluation, using self-reporting questionnaires and clinical findings, and quantitative evaluation, using laboratory measures of organ function and porphyrin levels, to evaluate the effectiveness of therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha C Balwani, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (15):
- United States (15):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Carolinas Medical Center and HealthCare System, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Balwani M, Naik H, Anderson KE, Bissell DM, Bloomer J, Bonkovsky HL, Phillips JD, Overbey JR, Wang B, Singal AK, Liu LU, Desnick RJ. Clinical, Biochemical, and Genetic Characterization of North American Patients With Erythropoietic Protoporphyria and X-linked Protoporphyria. JAMA Dermatol. 2017 Aug 1;153(8):789-796. doi: 10.1001/jamadermatol.2017.1557. PMID 28614581
- [Result] Saberi B, Naik H, Overbey JR, Erwin AL, Anderson KE, Bissell DM, Bonkovsky HL, Phillips JD, Wang B, K Singal A, M McGuire B, Desnick RJ, Balwani M. Hepatocellular Carcinoma in Acute Hepatic Porphyrias: Results from the Longitudinal Study of the U.S. Porphyrias Consortium. Hepatology. 2021 May;73(5):1736-1746. doi: 10.1002/hep.31460. Epub 2020 Dec 11. PMID 32681675
- [Result] Levy C, Naik H, Overbey J, Hedstrom K, Wang K, McDonough C, Freeman M, Keel SB, Erwin AL, Dickey AK, Leaf RK, Quigley J, Mazepa M, Wang B, Phillips J, Parker C, McGuire B, Kazamel M, Bonkovsky H, Rudnick S, Anderson KE, Moghe A, Thapar M, Saberi B, Wheeden K, Desnick R, Balwani M; Porphyrias Consortium of the Rare Diseases Clinical Research Network. Liver involvement in a large cohort of patients with erythropoietic protoporphyria or X-linked protoporphyria. Hepatol Commun. 2025 Feb 19;9(3):e0657. doi: 10.1097/HC9.0000000000000657. eCollection 2025 Mar 1. PMID 39969427
- [Derived] Bonkovsky HL, Maddukuri VC, Yazici C, Anderson KE, Bissell DM, Bloomer JR, Phillips JD, Naik H, Peter I, Baillargeon G, Bossi K, Gandolfo L, Light C, Bishop D, Desnick RJ. Acute porphyrias in the USA: features of 108 subjects from porphyrias consortium. Am J Med. 2014 Dec;127(12):1233-41. doi: 10.1016/j.amjmed.2014.06.036. Epub 2014 Jul 10. PMID 25016127
- See also: Website for the Rare Diseases Clinical Research Network (RDCRN) Porphyrias Consortium (PC — https://www.rarediseasesnetwork.org/cms/porphyrias